CLINICAL TRIAL: NCT00924846
Title: High-Frequency Oscillatory Ventilation Associated With Inhaled Nitric Oxide in Children: Randomized, Crossover Study
Brief Title: High-Frequency Oscillatory Ventilation Associated With Inhaled Nitric Oxide in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: José Roberto Fioretto, UNESP-Botucatu Medical School
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: upeclin/HC/FMB-Unesp-26
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Last update posted 2009-06-22 (Estimated); Status verified 2009-06

CONDITIONS: Acute Hypoxemic Respiratory Failure
Keywords: high frequency oscillatory ventilation; respiratory failure; children; inhaled nitric oxide
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- HFOV plus iNO (Active Comparator): HFOV plus iNO: high frequency oscillatory ventilation plus inhaled nitric oxide
  Interventions: Procedure: High frequency oscillatory ventilation
- CMV plus iNO (Active Comparator): CMV (conventional mechanical ventilation) iNO (inhaled nitric oxide)
  Interventions: Procedure: High frequency oscillatory ventilation

INTERVENTIONS:
Procedure: High frequency oscillatory ventilation — Mechanical ventilation as high frequency oscillatory ventilation for 8h periods
  Other Names: HFOV

SUMMARY:
Background/Objectives: Acute hypoxemic respiratory failure (AHRF) is a frequent cause of pediatric ICU admission. Early treatment with inhaled nitric oxide (iNO) plus conventional mechanical ventilation (CMV) improves oxygenation, responsiveness being significantly influenced by alveolar recruitment level. High-frequency oscillatory ventilation (HFV) is conceptually very attractive as constant mean airway pressure optimizes lung recruitment; this could maximize iNO effects.

Aims: To analyze the effects of HFV on oxygenation indexes in AHRF children under CMV and iNO.

Methods: Children with AHRF (oxygenation index ≥10) aged between one month and 14 years under CMV with PEEP≥10cmH2O and 5ppm iNO for 1h were randomly assigned to CMV (CMVG, n=12) or HFV (HFVG, n=12) in a crossover design. Children with chronic cardiac or pulmonary diseases were excluded. Patients were kept under one of the two ventilation modes for 8h, crossing to the other for 8h, and then back again to complete 24h observation. Blood gas analysis, oxygenation indexes, and hemodynamic variables were recorded at enrollment (Tind), 1h after iNO start and then every 4h (T4h etc). The Mann-Whitney U test compared group ages and PRISM scores, and the Fisher test genders. Moments and groups were compared by repeated measure analysis for independent groups. Significance was considered at p<0.05.

DETAILED DESCRIPTION:
Acute hypoxemic respiratory failure (AHRF) is a frequent cause of admission and complicates evolution of critically ill children. Mortality rate is still high, mainly when acute respiratory distress syndrome (ARDS) evolves.

Clinical management of AHRF is essentially supportive and includes control of underlying infections, fluid balance and hemodynamic status, nutritional support, and optimized protective mechanical ventilation4,5,6. Ventilatory strategies should be directed at minimizing ventilator-induced lung injury (VILI), eliminating oxygen toxicity, and controlling lung inflammation. Also, when hypoxemia persists, additional treatments may be implemented, such as inhaled nitric oxide (iNO)and high-frequency oscillatory ventilation (HFOV).

Recently, we have demonstrated that early treatment with iNO associated with protective conventional mechanical ventilation (CMV) causes acute and sustained improvement in oxygenation, with earlier reduction in ventilator settings that are associated with a high risk of VILI and oxygen toxicity; this might contribute to reducing the mortality rate in children with ARDS.

However, many studies have given no value to iNO therapy because of a lack of impact on mortality rate. Despite this, it should be considered that the improvement in oxygenation promoted by NO inhalation may be useful as rescue therapy. Also, it is known that responsiveness to iNO can be significantly influenced by applying sufficient positive and expiratory pressure (PEEP), as this seems to recruit additional alveoli for gas exchange. In this sense, HFOV is very attractive as the application of a constant mean airway pressure maintains an "open lung" and optimizes lung recruitment; this could maximize iNO effects.

Two experimental studies have shown increased iNO effects when the gas was used together with HFOV. In ARDS adults, Authors studied this association and demonstrated improvement in oxygenation with significant reduction in FiO2, probably due to the degree of alveolar recruitment during HFOV which may increase the amount of alveolar/capillary interface available for iNO to act upon.

In pediatrics, there is one study combining iNO and HFOV in newborn babies with severe persistent pulmonary hypertension which concluded that the association is often more successful than each treatment alone23. After neonatal period, a retrospective (post hoc) data analysis from a multicenter, randomized controlled trial on the effects of iNO in the treatment of AHRF concluded that the combination of HFOV with iNO causes greater improvement in oxygenation than either treatment strategy alone.

Therefore, the question about the potential role of the association between iNO therapy and HFOV in AHRF children is still open and remains to be defined. Our hypothesis is the association between early iNO treatment and HFOV improves oxygenation more consistently and for longer time than the association of the gas with protective conventional mechanical ventilation.

The aim of this study was to analyze the effects of HFOV on oxygenation indexes in AHRF children under CMV and iNO therapy.

ELIGIBILITY:
Inclusion Criteria:

* Children with AHRF (oxygenation index ≥ 10) aged between one month and 14 years under CMV with PEEP ≥ 10 cmH2O and 5 ppm iNO for 1 hour.

Exclusion Criteria:

* Children with chronic cardiac or pulmonary diseases.

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2005-04; Primary Completion 2008-04 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Oxygenation indexes | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jose R Fioretto, MD, PhD, Study Chair — UNESP-Botucatu Medical School
Locations (1):
- UNESP-Botucatu Medical School, Botucatu, São Paulo, Brazil